CLINICAL TRIAL: NCT02055898
Title: Slow-wave Sleep and Daytime Functioning in Chronic Fatigue Syndrome: Effects of Sodium Oxybate
Brief Title: SWS And Daytime Functioning in Chronic FatiguE Syndrome (SAFFE)
Acronym: SAFFE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: SAFFE2012; 2012-002969-35 (EudraCT Number)
Record Dates: First submitted 2013-12-13; First posted 2014-02-05 (Estimated); Results first posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-10

CONDITIONS: Chronic Fatigue Syndrome
Keywords: Chronic fatigue syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Sodium Oxybate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo first, then sodium oxybate (Experimental): Subjects received a single dose of placebo comparator (fresh potable water) at bedtime on 4 nights during an inpatient stay of 5 days in the research centre. This was followed by an interval of at least 2 weeks. They were then admitted again and received a single dose of sodium oxybate (3.0g as liquid) at bedtime for 4 nights
  Interventions: Drug: Sodium Oxybate; Other: placebo (fresh potable water)
- Sodium oxybate first, then placebo (Experimental): Subjects received a single dose of sodium oxybate (3.0g as liquid) at bedtime on 4 nights during an inpatient stay of 5 days in the research centre. This was followed by an interval of at least 2 weeks. They were then admitted again and received a single dose of placebo comparator (fresh potable water) at bedtime for 4 nights
  Interventions: Drug: Sodium Oxybate; Other: placebo (fresh potable water)

INTERVENTIONS:
Drug: Sodium Oxybate
  Other Names: Xyrem
Other: placebo (fresh potable water)

SUMMARY:
The investigators wish to investigate whether enhancement of SWS, which is seen after a drug called sodium oxybate, reduces the impact of sleep disruption in CFS on daytime function, specifically sleepiness and mental performance. This is a safe and well-tolerated drug that is licensed for excessive daytime sleepiness (EDS) and cataplexy associated with narcolepsy.

The investigators will study 12 patients diagnosed with CFS using international diagnostic guidelines. The investigators will record overnight sleep with EEG (brainwave) measurement on the 1st and 4th nights of a 4 night period during which sodium oxybate and placebo will be taken nightly, and the investigators will measure next-day sleepiness, mental performance and fatigue, and compare drug and placebo nights.

DETAILED DESCRIPTION:
Chronic fatigue syndrome (CFS), characterised by chronic disabling fatigue, sleep impairment and other symptoms, is associated with neither a currently identifiable disease process nor major psychiatric illness, and has an estimated prevalence in primary care of 1-2%. Sleep impairment is common in nearly everyone with CFS, with both daytime sleepiness and unrefreshing nighttime sleep reported, and consequent impact on daytime function. It may be that fundamental regulatory processes that control sleep are disturbed in CFS, leading to different effects on sleep and daytime symptoms depending on the subject's prior sleep, daytime routine, medication and other factors. The investigators contacts with patient groups have indicated that patients are generally confident that on days when their sleep is better they perform better in the day. There is growing evidence that deep, slow wave sleep (SWS) is altered in CFS, and this may suggest impairment of build up of sleep pressure during the day.

ELIGIBILITY:
Inclusion criteria

* Meeting criteria for CFS according to both the revised CDC (Fukuda 5) and Canadian diagnostic systems.
* Aged 25-65.
* Good grasp of the English language.

Exclusion criteria

* Taking any of the following medication: opioids, tramadol, phenytoin, valproate, ethosuximide, benzodiazepines, zolpidem, zopiclone, zaleplon, antidepressant except <30mg amitriptyline, or any other medications likely to interact with sodium oxybate or with sleep in the opinion of the investigators.
* Current major psychiatric disorder.
* Unusual sleep schedule; (bedtime routines that fall outside 9 p.m. to 10 a.m.; usual time in bed > 12 hours).
* Pregnancy, lactation or being female and not using reliable contraception.
* Relevant abnormal clinical findings at screening visit.
* Taken alcohol in the 24 hours before each study visit or drugs of abuse in the week before each study visit

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Nutt, DM FRCPsych, Principal Investigator — Imperial College London
Locations (1):
- Wellcome CRF, Imperial College, Hammersmith Campus, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Then Sodium Oxybate: 7 patients with chronic fatigue syndrome
- Sodium Oxybate Then Placebo: 6 patients with chronic fatigue syndrome
Period: First Intervention (5 Days)
Arm/Group | Placebo Then Sodium Oxybate | Sodium Oxybate Then Placebo
Started | 7 | 6
Completed | 5 | 5
Not Completed | 2 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout (at Least 14 Days)
Arm/Group | Placebo Then Sodium Oxybate | Sodium Oxybate Then Placebo
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Second Intervention (5 Days)
Arm/Group | Placebo Then Sodium Oxybate | Sodium Oxybate Then Placebo
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo First Then Sodium Oxybate: 7 Patients who meet criteria for CFS according to both the revised CDC (Fukuda 5) and Canadian diagnostic systems.
- Sodium Oxybate First Then Placebo: 6 Patients who meet criteria for CFS according to both the revised CDC (Fukuda 5) and Canadian diagnostic systems.
- Total: Total of all reporting groups
Arm/Group | Placebo First Then Sodium Oxybate | Sodium Oxybate First Then Placebo | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United Kingdom | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: EEG Slow Wave Activity During Sleep
Description: Total power in 0.5-4Hz band in microvolts squared per Hertz (uV^2/Hz)
Time Frame: night 1
Population: All participants who completed the study and whose recordings were adequate
Measure: Mean (Standard Error); unit: uV^2/Hz
Groups:
- Sodium Oxybate: All participants who completed the study and whose recordings were adequate, during the sodium oxybate period
- Placebo: All participants who completed the study, and whose recordings were adequate, during the placebo period
Arm/Group | Sodium Oxybate | Placebo
Number analyzed (Participants) | 9 | 9
uV^2/Hz | 0.00002653 (0.00000406) | 0.00002257 (0.00000339)

2. Primary Outcome: EEG Slow Wave Activity During Sleep
Description: Total power in 0.5-4Hz band in microvolts squared per Hertz (uV^2/Hz)
Time Frame: night 4
Population: All participants who completed the study and whose recordings were adequate
Measure: Mean (Standard Error); unit: uV^2/Hz
Arm/Group | Sodium Oxybate | Placebo
Number analyzed (Participants) | 9 | 9
uV^2/Hz | 0.00003051 (0.00000492) | 0.00001759 (0.00000225)

3. Primary Outcome: Daytime Sleepiness
Description: time to fall asleep in minutes
Time Frame: Day 2
Population: All participants who completed the study and whose recordings were adequate
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Sodium Oxybate | Placebo
Number analyzed (Participants) | 10 | 10
minutes | 16.95 (0.773) | 15.3 (1.35)

4. Primary Outcome: Daytime Sleepiness
Description: time to fall asleep in minutes
Time Frame: Day 5
Population: All participants who completed the study
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Sodium Oxybate | Placebo
Number analyzed (Participants) | 10 | 10
minutes | 17.9 (0.9) | 17.2 (1.2)

ADVERSE EVENTS:
Time Frame: 2 months
Groups:
- Placebo: All participants who received at least one dose of placebo
- Sodium Oxybate: All participants who received at least one dose of sodium oxybate
Arm/Group | Placebo | Sodium Oxybate
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 6/12 | 5/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | Sodium Oxybate (N=11)
Obstructive sleep apnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
itchy skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) — mild itchiness
painful legs at night (General disorders) | 1 (1) | 0 (0)
hay fever (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Indigestion/upset stomach (Gastrointestinal disorders) | 0 (0) | 4 (4) — including mild nausea
central sleep apneas (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — as recorded with overnight polysomnography
headache (General disorders) | 0 (0) | 2 (2)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
unsteadiness (General disorders) | 0 (0) | 1 (1)
feels confused on waking (General disorders) | 0 (0) | 2 (2) — Brief period of disorientation on waking

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes